CLINICAL TRIAL: NCT03464006
Title: Online Support for Outpatient Peripheral Arterial Disease Self-management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: Reliq Health Technologies Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAD Management
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a single centre, randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Support Module (Experimental): Patients in the online support module group will receive a tablet which has the developed peripheral arterial disease platform installed on it. The platform helps the patient to monitor factors related to their peripheral arterial disease such as exercise, smoking, and diet and helps them to track and modify these behaviours.
  Interventions: Other: Online Support Module
- Standard of Care (Active Comparator): Patients in this arm will receive the standard of care as provided by the institution.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Online Support Module — The online support module is a computer software program which helps patients monitor factors related to their peripheral artery disease
  Arms: Online Support Module
Other: Standard of Care — The normal care that patients receive at the institution.
  Arms: Standard of Care

SUMMARY:
This study looks to examine whether an online patient tool to monitor factors affecting patients peripheral artery disease can lead to improvements in patients' disease and slow its progression.

DETAILED DESCRIPTION:
The objective of this project is to implement a program involving a new online patient-centred approach to assist in peripheral arterial disease (PAD) self-management in home and work environments, in collaboration with patient circles of care (patients, care-givers, physicians, and allied healthcare professionals). This program involves online modules tailored to the needs of specific patients and diseases, oriented to education, training, monitoring, and continuing support for lifestyle changes (smoking cessation, exercise, healthy diets, weight loss, etc.) and psycho-social needs such as social isolation and loneliness. The investigators have tested an online desk-top version for over 30 out-patients with PAD at St. Michael's Hospital in Toronto. The investigators propose to test its ability for improved outcomes and healthcare quality of life through a multi-centre randomized controlled trial for PAD and a frequently co-occurring chronic illness, high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* diagnosed with peripheral artery disease (ABI<0.9)

Exclusion Criteria:

* unable to communicate in English
* unwilling to participate
* patients with dementia or other cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Ankle Brachial Index | 1 year
  The ankle brachial index will be measured to determine peripheral artery disease status and progression.

SECONDARY OUTCOMES:
Blood Pressure | 1 year
  Patient blood pressure.
Health Related Quality of Life | 1 year
  Quality of life measured using the EuroQol-5D (EQ-5D). The EQ-5D provides a variety of health states which can then be converted to an index score ranging from 0-1.0, with 0 indicating a poorer health state and 1.0 representing a better health state.
Diabetes Status | 1 year
  Diabetes status measured by hemoglobin A1C
Vascular Health | 1 year
  Measured using LDL, HDL, and total cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Stacey, DS, Principal Investigator — McMast

IPD SHARING:
Plan to Share IPD: No
There is no plan to share patient level data.